CLINICAL TRIAL: NCT01174134
Title: The Effects of Study Products Containing Varying Quantities of Docosahexaenoic Acid (DHA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Carol Berseth, M.D., Mead Johnson Nutrition
Other Study IDs: 3375-1
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Levels of DHA in the Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk-based beverage w/out DHA (Placebo Comparator)
  Interventions: Other: Nutritional beverage
- Milk-based beverage with DHA (Experimental)
  Interventions: Other: Nutritional beverage
- Milk-based beverage containing DHA at a higher level (Experimental)
  Interventions: Other: Nutritional beverage

INTERVENTIONS:
Other: Nutritional beverage

SUMMARY:
The clinical trial will provide a milk-based drink with constant amounts of nutrients but differing amount of Docosahexaenoic Acid (DHA).

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 to 36 months of age
* Participant's current weight and height within the 10th to 90th percentiles
* Parent/caregiver reports that participant consumes milk or a milk-based beverage on a daily basis
* Participant lives at home with parent(s) or other family member(s)
* Signed informed consent and authorization obtained to use and or disclose Protected Health Information (PHI)

Exclusion Criteria:

* Participant who is receiving any breast milk at time of randomization
* Participant with an active infection.
* Participant with a history of underlying disease, chronic disease, or congenital malformation which in the opinion of the Investigator is likely to interfere with the evaluation of the participant.
* Known or suspected intolerance to cow's milk protein
* Participant diagnosed with diabetes
* Participant is from a multiple birth and the sibling(s) are still living
* Participant with a sibling that has participated in this study.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2006-07; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Blood lipid levels of Docosahexaenoic Acid (DHA) at enrollment and after two months, assessment of usual DHA intake, and product acceptability and use

SECONDARY OUTCOMES:
Growth
Determination of nutrient status, including iron and vitamin D status
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Susan Carlson, Ph.D., Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Kansas City, Kansas, United States